CLINICAL TRIAL: NCT06837337
Title: The Effect of Turkish Music
Brief Title: The Effect of Turkish Music on Pain and Anxiety During Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinop University (Other)
Collaborators: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 03-2023/18
Record Dates: First submitted 2025-01-17; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Childbirth; Pain; Anxiety
Keywords: Nursing Caries; childbirth pain; music; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders; Labor Pain

STUDY DESIGN:
Intervention Model Description: Randomized control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- music group (Experimental)
  Interventions: Other: Music intervention
- control group (No Intervention)

INTERVENTIONS:
Other: Music intervention — Music intervention
  Arms: music group

SUMMARY:
Nurses and midwives stand at the forefront during childbirth; their expertise in using natural pain relief techniques not only lessens the sensation of labor pain but also helps in calming the nerves of expectant mothers. These techniques are not only safe and easy to use but also kind on the pocket and devoid of any adverse effects. Such methods can make childbirth experiences as positive and comfortable as possible. Research has delved deeper into how music shaped by cultural tastes can significantly affect individuals, leading to a closer examination of how Turkish tunes influence discomfort and nervousness during labor. The goal of this research was to explore how Turkish melodies impact pain and anxiety feelings among women going through childbirth for the first time.

ELIGIBILITY:
Inclusion Criteria:

* primigravida women with term pregnancies (38-40 weeks) in the early active phase of labor
* cervical dilatation between 4 and 6 cm

Exclusion Criteria:

* Women who used narcotic analgesics or sedatives during labor
* listened to music during childbirth
* underwent induction
* delivered via cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Angle Labor Pain Questionnaire | Approximately one hour after admission to the delivery room, change from the initial pain level in 30 minutes. Scores of Angle Labor Pain Questionnaire ranged from 0 to 220, with higher values indicating greater pain intensity.
  Pain Level by Angle Labor Pain Questionnaire.
Visual Analog Scale (VAS) | Approximately one hour after admission to the delivery room, change from the initial pain level in 30 minutes. VAS is a 10 cm line used to measure perceived pain intensity, with endpoints labeled "No Pain" and "Worst Pain Imaginable."
  Pain Level by Visual Analog Scale (VAS)
The State Anxiety Scale (SAS) | Approximately one hour after admission to the delivery room, change from the initial anxiety level in 30 minutes. The total scores range from 20 to 80, with higher scores indicating greater anxiety.
  The State Anxiety Scale (SAS) measures anxiety as a temporary emotional state.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinop University, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing is not considered appropriate until the article has completed its journal process and is published.

REFERENCES:
- [Background] Guo H, Que M, Shen J, Nie Q, Chen Y, Huang Q, Jin A. Effect of Music Therapy Combined with Free Position Delivery on Labor Pain and Birth Outcomes. Appl Bionics Biomech. 2022 May 11;2022:8963656. doi: 10.1155/2022/8963656. eCollection 2022. PMID 35600844